CLINICAL TRIAL: NCT04402346
Title: Radiofrequency-assisted Transection of the Pancreas vs Stapler. A Phase III Randomized Clinical Trial.
Brief Title: Radiofrequency-assisted Transection of the Pancreas vs Stapler
Acronym: TRANSPAIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Sanchez Velazquez (Other)
Responsible Party: Sponsor-Investigator, Patricia Sanchez Velazquez, Principal Investigator, Hospital del Mar
Organization: Hospital del Mar (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMar_RF_transection_pancreas
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Pancreas; Fistula
Keywords: Pancreas fistula; Distal pancreatectomy; Radiofrequency
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency-assisted (Experimental)
  Interventions: Procedure: Radiofrequency-assisted pancreas transection
- Stapler (Active Comparator)
  Interventions: Procedure: Stapler assisted pancreas transection

INTERVENTIONS:
Procedure: Radiofrequency-assisted pancreas transection — Transection of the pancreas in distal pancreatectomy by applying a radio frequency device
  Arms: Radiofrequency-assisted
Procedure: Stapler assisted pancreas transection — Transection of the pancreas in distal pancreatectomy by applying a stapler device with/without seamguard
  Arms: Stapler

SUMMARY:
Main objective: The main end-point of this study is to compare in a randomized clinical trial that radiofrequency-assisted pancreas transection (RF) reduces the incidence of postoperative pancreatic fistula (POPF) compared to the classical method of transection (stapler). As secondary end-points, other clinical and demographic variables of the patients will be evaluated (sex, age, ASA classification, consistency of the pancreas, as well as the type of procedure, open or laparoscopic surgery, estimated intraoperative bleeding, pancreatic duct size, duration of intervention, type of tumor and quality of lymphatic resection). Methodology: Phase III prospective multicenter study in patients undergoing distal pancreatectomy for any origin. All consecutive patients who undergo a distal pancreatectomy for any cause in a multicenter setting will be included. A simple randomization of the participants to the RFA group or to the control group (stapler) will be carried out. The incidence of pancreatic fistula will be assessed as main variable; predictive multivariable models with multiple regression for quantitative variables, logistic regression for categorical variables and Cox regression for survival analyzes. In addition to histological study, molecular analysis of resection specimen and clinical and radiological follow-up with volumetry of necrosis in the area of post-pancreatectomy transection will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Solid or cystic, benign or malign pancreas neoplasms.
* Patients undergoing a distal pancreatectomy, i.e pancreas transection beyond > 2 cm from the SMV (assessed by computer tomography or RM) with or without splenectomy
* Both open and laparoscopic approaches are valid.

Exclusion Criteria:

* Patients who required a pancreatectomy with transection at the level of the neck.
* Non-intervention group: only stapler transection will be accepted, other pancreatic transection methods will be excluded.
* Patients ASA≥IV
* Absence of informed consent
* Underage (<18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pancreas fistula | 90 days follow-up
  Defined by the updated 2016 ISGPF definition

SECONDARY OUTCOMES:
In-hospital Mortality | In-Hospital (30 days)
  30 days
Morbidity | 90 days follow-up
  In terms of Clavien-Dindo and CCI classification

CONTACTS AND LOCATIONS:
Locations (1):
- Parc de Salut Mar de Barcelona- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Velazquez P, Pueyo-Periz E, Alamo JM, Suarez Artacho G, Gomez Bravo MA, Marcello M, Vicente E, Quijano Y, Ferri V, Caruso R, Dorcaratto D, Sabater L, Gonzalez Chavez P, Noguera J, Navarro Gonzalo A, Bellido-Luque J, Tellez-Marques C, Ielpo B, Burdio F. Radiofrequency-assisted transection of the pancreas versus stapler in distal pancreatectomy: study protocol for a multicentric randomised clinical trial (TRANSPAIRE). BMJ Open. 2022 Nov 4;12(11):e062873. doi: 10.1136/bmjopen-2022-062873. PMID 36332946